CLINICAL TRIAL: NCT06513546
Title: A Multi-centre, Phase 1/2, Randomised, Double-blind, Placebo Controlled Study With an Optional Open-label Extension to Evaluate the Safety, Tolerability, Efficacy, and Pharmacodynamics of PLL001 for the Treatment of ALS
Brief Title: A Study to Evaluate the Safety, Efficacy, and Pharmacodynamics of PLL001 in ALS Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PLL TX AUSTRALIA PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLL001-101
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Acetates; Butyrates; Lactic Acid; Propionates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLL001 dose 5x (Experimental): PLL001 lowest dose (Poly-l-Lysine conjugates with acetate, butirate, lactate, propionate) daily subcutaneous injections
  Interventions: Drug: PLL001 or placebo daily subcutaneous injections
- PLL001 dose 10x (Experimental): PLL001 highest dose (Poly-l-Lysine conjugates with acetate, butirate, lactate, propionate) daily subcutaneous injections
  Interventions: Drug: PLL001 or placebo daily subcutaneous injections
- placebo (Placebo Comparator): Saline daily subcutaneous injections
  Interventions: Drug: PLL001 or placebo daily subcutaneous injections

INTERVENTIONS:
Drug: PLL001 or placebo daily subcutaneous injections — PLL001 consists of the combination of 4 drug substances (DS) each being a linear poly-lysine flexible backbone with an average length of 70 L-lysines linked with 10% of conjugated side chains all being small chain fatty acids (SCFAs) (acetate, butyrate, lactate and propionate). The remaining 90% of the lysine residues are present as bromide salt. PLL001 DP is presented as 20 mL vials containing 16 mL of a sterilised solution for SC injection with the following formula (5× concentration)
  Other Names: Poly-L-lysine conjugates with acetate, butyrate, lactate, propionate

SUMMARY:
FIH, Phase 1/2, multi-centre, randomised, double-blind, placebo controlled study with an optional open-label dosing extension to assess the safety, tolerability, efficacy, and Pharmacodynamics (PD) of single or multiple (up to 48 weeks QD) subcutaneous (SC) doses of PLL001 compared to placebo in subjects diagnosed with ALS.

DETAILED DESCRIPTION:
Part 1 (Single Ascending Dose A total of 12 subjects will be randomised to 1 of 3 dose level cohorts (4 subjects per cohort). In each cohort, subjects will be randomised at a ratio of 3:1 to receive a single SC dose of PLL001 or placebo in a double-blind manner. The safety data of placebo subjects will be pooled.

Subjects will be admitted to the unit on the day prior to dosing (Day -1) and will be administered in a double-blind manner PLL001 or placebo via SC injection in the morning on Day 1. Subjects will remain hospitalised for a minimum of 24 hours for safety evaluation and will be discharged in the morning on Day 2. Safety data will be collected daily up to Day 7 (End of Study [EOS]).

Subjects that have completed Part 1 of the study will be eligible for screening in Part 2.

Part 2 (Multiple Dose Expansion)

Up to 141 subjects will be randomised to 1 of 3 treatments groups (2 dose level groups of PLL001 and 1 group of placebo) at a ratio of 1:1:1 (40 subjects per treatment group plus 21 patients for drop-out replacements).

The first 21 subjects (ie, 7 subjects per treatment group) will be dosed initially and will be randomised to 1 of the 3 treatment groups at a ratio of 1:1:1. These first 21 subjects will be monitored for the first 14 days of QD dosing. Following review of the safety data by the SRC and in the absence of any clinically significant safety signals, the remaining subjects will be enrolled.

Patients under riluzole will be allowed to continue their riluzole treatment and will be stratified at randomisation in Part 2 to ensure comparable numbers between each treatment group. Patients will also be stratified at randomisation in Part 2 based on TRICALS' risk profile calculator score (https://tricals.shinyapps.io/risk-profile/) to ensure comparable patients' ALS profiles between each treatment group.

Subjects will self-administer or have carers administer PLL001 or placebo daily (QD) via 2 × SC injections of 1 mL in a double-blind manner.

Addmionsitrationbs will be on-site on the morning of Day 1 and will self-administer or have carers administer on all other dosing days stopping the day before the visit on Day 169 (±5 days). Subjects will be discharged after a 4-hour observation period post-administration on Day 1.

Efficacy, safety, and compliance data will be collected during site visits which will occur every 8 weeks on Day 57, 113 and 169 (±5 days) (plus on Day 15 for all treated subjects).

Safety and compliance data will be collected via tele contact weekly (±3 days) on the weeks subjects do not attend a site visit.

Part 3 (Open-label Extension)

Subjects that consent to with the optional open-label treatment will commence open-label treatment at the visit on Day 169 (±5 days) and continue daily self dosing (or carer-administered dosing) of PLL001 10× via 2 × SC injections of 1 mL for an additional 24 weeks (for a total of 48 weeks of treatment) stopping the day before the visit on Day 337 (±5 days).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age at the time of informed consent.
2. Diagnosed within the previous 1 year with laboratory-supported probable, clinically probable or definite ALS according to the World Federation of Neurology Revised El Escorial criteria.
3. Must have familial or sporadic ALS.
4. First ALS symptoms occurred no more than two (2) years prior to screening visit ALS disease duration from diagnosis no longer than 12 months at the Screening visit.
5. If treated with riluzole, edaravone or any other approved ALS medication, treated with a stable dose for at least 4 weeks prior to Day 1.
6. If documented, patient with an ALSFRS-R score progression between onset of the disease and Screening of > 0.3 per month, confirmed with an ALSFRS-R score progression of ≥ 1 point during a 12 week prior to randomisation.
7. Has a score of at least 26 overall, including a score of at least 3 on item #3 and at least 2 on each of the 12 ALSFRS-R individual component items at Screening and at least 2 on each of the 12 ALSFRS-R individual component items at randomisation.
8. Seated slow vital capacity (SVC) ≥ 50% of predicted value for gender, height, and age at screening.
9. Must be willing and able to comply with the requirements of the protocol and must be available to complete the study.
10. Must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Has dementia or significant neurological, psychiatric, systemic, or organic disease, uncontrolled or that may interfere with the conduct of the trial or its results.
2. Pregnant or nursing females.
3. History of drug/chemical/substance/alcohol abuse within the past 2 years prior to Screening, including cannabinoid therapies.
4. Significant symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within the past 2 weeks prior to study medication administration (at the discretion of the Investigator).
5. Mechanical ventilation via tracheostomy or dependence on non-invasive ventilation, (> 16 hours / day). (Lesser intermittent use of non-invasive ventilation eg, continuous positive airway pressure, non-invasive bi-level positive airway pressure or non-invasive volume ventilation is not an exclusion).
6. Patients positive for human immunodeficiency virus (HIV) antibody, hepatitis C antibody, or for hepatitis B virus surface antigen (HBsAg).
7. Sexually active females of childbearing potential and male subjects who are not practicing at least one method of hormonal or mechanical birth control with their partner during the study and for 90 days after the last dose of the study medication. Males and females who are not heterosexually active or who practice true abstinence are exempt from contraceptive requirements.
8. Experimental agent within 30 days or 5 half-lives, whichever is longer, prior to study drug administration (Part 1 only).
9. Any other condition which, in the opinion of the Investigator, precludes participation in the study.
10. Dependents of the Sponsor or Investigator.
11. Known allergy to the study drug and/or its constituents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Part 1: safety | 7 days
  AEs, change from Baseline in other safety parameters (metric values) Haemotology: Haemoglobin g/L; Haematocrit L/L; Red Blood Cells X10^12/L; White Blood Cells X10^9/L; Platelets X10^9/L; Neutrophils X10^9/L; Eosinophils X10^9/L; Lymphocytes X10^9/L; Monocytes X10^9/L; Basophils X10^9/L; Mean corpuscular volume fL Biochemistry: Sodium mmol/L; Potassium mmol/L; Phosphate mmol/L; Calcium mmol/L; Urea mmol/L; Uric Acid mmol/L; Creatinine umol/L; Glucose mmol/L; Protein g/L; Albumin g/L; Bilirubin umol/L; ALP U/L; AST U/L; ALT U/L; GGT U/L; LDH U/L Coagulation: Prothrombin time sec; APTT sec; International Normalised Ratio; Fibrinogen g/L Urinalysis: RBC x10^6/L; WBC x10^6/L
Part 2: efficacy of PLL001 compared to placebo after 8, 16, and 24 weeks of once daily (QD) treatment | 24 weeks
  Change from Baseline in ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised) scores. Minimum score of 0 and a maximum score of 48. Higher scores indicate better functional status and retained abilities. Specifically, a score of 48 represents the best functional status, while a score of 0 indicates the worst functional status
Part 2: survival after 8, 16, and 24 weeks of QD treatment for PLL001 compared to placebo | 24 weeks
  Survival

SECONDARY OUTCOMES:
Part 2: safety | 24 weeks
  AEs, change from Baseline in other safety parameters (metric values) Haemotology: Haemoglobin g/L; Haematocrit L/L; Red Blood Cells X10^12/L; White Blood Cells X10^9/L; Platelets X10^9/L; Neutrophils X10^9/L; Eosinophils X10^9/L; Lymphocytes X10^9/L; Monocytes X10^9/L; Basophils X10^9/L; Mean corpuscular volume fL Biochemistry: Sodium mmol/L; Potassium mmol/L; Phosphate mmol/L; Calcium mmol/L; Urea mmol/L; Uric Acid mmol/L; Creatinine umol/L; Glucose mmol/L; Protein g/L; Albumin g/L; Bilirubin umol/L; ALP U/L; AST U/L; ALT U/L; GGT U/L; LDH U/L Coagulation: Prothrombin time sec; APTT sec; International Normalised Ratio; Fibrinogen g/L Urinalysis: RBC x10^6/L; WBC x10^6/L
Part 2: efficacy over 24 weeks | 24 weeks
  Progression-free survival (PFS)
  * Quality of life based on ALSAQ-40 score (Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 questions)
  * Respiratory function regression on Slow Vital Capacity score (SVC)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Soulis, Study Director — Alithialifesciences
Locations (10):
- Australia (10):
  - Liverpool Hospital, Liverpool, New South Wales
  - Neuroscience Research Australia, Sydney, New South Wlaes
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Wesley Research Institute, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Alfred Health, Melbourne, Victoria
  - Calvary Health Care, Bethlehem, Melbourne, Victoria
  - Monash Medical Centre, Neuroscience Research, Melbourne, Victoria
  - The Perron Institute for Neurological and Translational Science, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No